CLINICAL TRIAL: NCT06762210
Title: The Effectiveness of AI Molar Mind for Smoking Cessation Through Dental Health Evaluation: Randomized Control Trial
Brief Title: The Effectiveness of AI Molar Mind for Smoking Cessation Through Dental Health Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, prof. Oral & Maxillofacial Surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Oral health assessment AI
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking cessation; oral health
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, single-blind clinical trial with two parallel arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI Molar Mind Group (Experimental): Participants receive a baseline oral health assessment using AI Molar Mind
  Interventions: Other: AI Molar Mind
- Control group (No Intervention): Participants receive standard smoking cessation care

INTERVENTIONS:
Other: AI Molar Mind — a baseline oral health assessment using AI Molar Mind, which analyzes intraoral images and self-reported oral health data.
  Arms: AI Molar Mind Group

SUMMARY:
Smoking cessation remains a significant public health challenge, with millions of individuals struggling to quit despite available interventions.

DETAILED DESCRIPTION:
Oral health deterioration is a well-documented consequence of smoking, including periodontal disease, tooth discoloration, and oral cancer. Recent advancements in artificial intelligence (AI) have led to the development of AI Molar Mind, a digital tool designed to assess oral health and provide personalized feedback to motivate behavioral change. This study aims to evaluate the efficacy of AI Molar Mind in aiding smoking cessation by leveraging oral health evaluations as a motivational tool.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* smoke ≥5 cigarettes per day
* motivated to quit smoking,
* have access to a smartphone or computer

Exclusion Criteria:

* Pregnant women
* individuals with severe psychiatric conditions
* those already using other smoking cessation therapies.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
smoking cessation indicator | base line, 6-month post smoking cessation
  Biochemically verified smoking cessation at 6 months (measured by exhaled carbon monoxide levels <6 ppm).

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Mohamed, PhD, Principal Investigator — Fayoum University
Locations (1):
- faculty of Dentistry, Fayoum University, Fayoum, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oya-Watanabe Y, Inagaki K, Nimi T, Yamamoto Y, Tanabe T, Okai M, Segawa N, Watanabe T, Uchibori N, Koide T, Inukai J, Yuasa H, Mitani A, Nagao T, Fukui M, Hinode D. Attitudes toward smoking cessation according to smoking status among dentists in the Aichi Dental Association in Japan. Tob Induc Dis. 2024 Aug 6;22. doi: 10.18332/tid/191290. eCollection 2024. PMID 39109252
- [Background] Herpich TL, Mendes EM, Roxo-Goncalves M, Katz N, Almeida JD, Martins MD, Romanini J, Carrard VC. Impact of an educational intervention regarding tobacco counseling on dentists and dental students. Braz Oral Res. 2024 Nov 8;38:e102. doi: 10.1590/1807-3107bor-2024.vol38.0102. eCollection 2024. PMID 39536203